CLINICAL TRIAL: NCT00785590
Title: Dermatological Evaluation of the Photo Irritation and Photo Sensitivity Potential for Dermacyd PH_DETINLYN (Lactic Acid) Sweet Flower.
Brief Title: Dermacyd PH_DETINLYN (Lactic Acid) Sweet Flower - Photo Evaluation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_04300
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

ARMS (1):
- 1 (Experimental): Dermacyd PH_DETINLYN (Lactic Acid)
  Interventions: Drug: Dermacyd PH_DETINLYN (Lactic Acid)

INTERVENTIONS:
Drug: Dermacyd PH_DETINLYN (Lactic Acid)

SUMMARY:
To demonstrate the absence of photoirritation and photosensitization potential of the product Dermacyd PHDETINLYN Sweet Flower.

ELIGIBILITY:
Inclusion criteria:

* Phototype Skin II and III;
* Integral skin test in the region;
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time for medical evaluations and for application of occlusion;

Exclusion criteria:

* Lactation or gestation
* Use of Antiinflammatory and/or immunosuppression drugs 15 days before the selection;
* Diseases which can cause immunity decrease, such as HIV, diabetes;
* Use of drug photosensitizer;
* History of sensitivity or irritation for topic products;
* Active cutaneous disease which can change the study results;
* History of photodermatosis active;
* Family or personal antecedent of cutaneous photoinduced neoplasias;
* Presence of a precursor lesion of cutaneous neoplasia, such as nevus melanocyte and queratoses actinium;
* Intense solar exposure in the study area;
* Use of new drugs or cosmetics during the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The photo irritation test and the photosensitivity will be measured using UVA irradiation and evaluated according International Contact Dermatitis Research Group (ICDRG) scale | Throughout the study
The sensibility will be evaluated according to the skin type. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil